CLINICAL TRIAL: NCT02192762
Title: A Pilot Study of Withdrawal Regulation Training vs. Relaxation Training for Smoking Cessation (Withdrawal Exposure With Withdrawal Regulation Training for Smoking Cessation)
Brief Title: Withdrawal Exposure With Withdrawal Regulation Training for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Peter Hendricks, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F110601002
Record Dates: First submitted 2014-04-10; First posted 2014-07-17 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Withdrawal regulation training (Experimental): Withdrawal coping skills
  Interventions: Behavioral: Withdrawal regulation training
- Relaxation training (Active Comparator): Relaxation skills instruction
  Interventions: Behavioral: Relaxation training

INTERVENTIONS:
Behavioral: Withdrawal regulation training — Withdrawal coping skills
  Arms: Withdrawal regulation training
Behavioral: Relaxation training — Relaxation skills instruction
  Arms: Relaxation training

SUMMARY:
This is a pilot study of a withdrawal regulation training program compared to relaxation training for individuals that are interested in smoking cessation.

DETAILED DESCRIPTION:
Participants will be recruited through newspaper and internet advertisements, advertisements on public transportation, community centers and community based organizations. All recruitment materials will contain a toll-free telephone number with 24-hour voice mail. The first contact with potential participant will be by telephone interview to assess for eligibility of participant. Participants who meet eligibility criteria will be invited to an orientation meeting where a breath carbon monoxide sample will be obtained. Women participant of childbearing potential will have a pregnancy test administered.

Participants will be randomized to one of two conditions: Early Withdrawal Exposure + Withdrawal Relaxation Training (E+WT) or Relaxation Training (RT) control. The E+WT condition will consist of the development, application, modification, and repeated practice of individualized withdrawal regulation for behavioral and cognitive strategies. the RT condition will control for the therapeutic contact received by those in the E+WT condition and will consist of the development, application, modification, and repeated practice of individualized relaxation techniques (e.g. breathing exercises, imagery).

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 19 years of age
* Reports smoking at least 10 cigarettes per day
* Must have expired breath carbon monoxide reading of at least eight parts per million
* Report the intention to quit smoking
* Reside in the Birmingham area with no plan to relocate outside of the area in the next six months
* Have access to a telephone for scheduling follow up assessments

Exclusion Criteria:

* Inability to speak English
* Presence of a condition that contraindicates use of transdermal nicotine patch (i.e. angina pectoris, arrhythmia, recent myocardial infarction, allergies to adhesives, serious skin disorders, and current pregnancy or breast feeding)
* Presence of conditions that might interfere with compliance with protocol or greatly complicate treatment (i.e. current alcohol or other substance dependence, dementia, psychosis, schizophrenia, bipolar disorder, suicidal or homicidal ideation, and any disease acutely life-threatening or so severe that the participant cannot comply with the protocol)
* Concurrent participation in a formal treatment program for smoking cessation
* Current use of any pharmacotherapy for smoking cessation

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Biochemically verified smoking abstinence | 2 months after end-of-treatment
  Smoking abstinence will be determined by self-report and confirmed via breath carbon monoxide (CO) analysis. Self-report of no smoking over the past 7 days (7-day point prevalence abstinence) and a CO value of less than 8 parts per million will be indicative of smoking abstinence. Self-report of any smoking over the past 7 days and/or CO values of 8 or greater will be indicative of cigarette use.
Biochemically-verified smoking abstinence | 3 months after end-of-treatment
  Smoking abstinence will be determined by self-report and confirmed via breath carbon monoxide (CO) analysis. Self-report of no smoking over the past 7 days (7-day point prevalence abstinence) and a CO value of less than 8 parts per million will be indicative of smoking abstinence. Self-report of any smoking over the past 7 days and/or CO values of 8 or greater will be indicative of cigarette use.

SECONDARY OUTCOMES:
Withdrawal symptoms | 2 months after end-of-treatment
  Withdrawal symptoms will be measured via self-report with the Wisconsin Smoking Withdrawal Scale (WSWS), a reliable and valid instrument of smoking withdrawal symptomatology.
Withdrawal symptoms | 3 months after end-of-treament
  Withdrawal symptoms will be measured via self-report with the Wisconsin Smoking Withdrawal Scale (WSWS), a reliable and valid instrument of smoking withdrawal symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Hendricks, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States